CLINICAL TRIAL: NCT01865422
Title: French Linguistic and Metric Validations of Parent-proxy QOL Chronic Cough Specific Questionnaire (PC-QOL)
Acronym: PC-QOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012-A01548-35; 2012-42 (Other: AP HM)
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chronic cough (Experimental)
  Interventions: Other: parent-proxy QoL chronic cough specific questionnaire (PC-QOL)

INTERVENTIONS:
Other: parent-proxy QoL chronic cough specific questionnaire (PC-QOL)

SUMMARY:
Cough is one of the most common reasons for consultation. Even if cough is a non-specific symptom, it can be the first sign of a chronic pathology. Several studies have demonstrated that chronic cough causes quality-of-life (QoL) impairment. Physicians' incapability to evaluate cough impact and patients' QoL has been documented. Therefore, a parent-proxy QoL chronic cough specific questionnaire (PC-QOL) has been developed and validated by Chang A. B.

Objective : The aim of the study is to validate the French version of the PC-QoL, a parent-proxy QoL chronic cough specific questionnaire.

Methods : Linguistic validation will be performed using backward/forward translation guidelines, and cognitive debriefing by 10 parents. Psychometric validation will be tested in 150 patients. Inclusion criteria are: patients with a diagnosis of chronic cough (> 4 weeks); 18 years of age or younger; all etiologies excepting cystic fibrosis. Informed consent from parents will be obtained. At enrollement, each parent will fulfill the PC-QOL questionnaire and two cough-related measures (visual analogue score, verbal category descriptive). Clinical data (medical history, physical examination) will be collected. Children QoL will be assessed using VSPA, Kidscreen and Qualin questionnaires. For assessing reproductibility and sensitivity to change, parents will be retested 7 and 21 days later. Content validity, construct's validity, external validity and instrument's reliability will be explored.

ELIGIBILITY:
Inclusion Criteria:

Old under age 18

* Male or feminine
* Reached(Affected) by chronic cough ( more than 4 weeks), any confused(merged) étiologie
* Affiliated to a national insurance scheme
* Having given freely their written consent having been informed about the purpose, about the progress and about the incurred potential risks

Exclusion Criteria:

Patients of whom the parents(relatives) are incapable to understand(include) the purpose and the conditions of realization of the study, incapable to give their consent

* Patient whose membership(support) to the protocol is improbable according to the investigator
* Patient participant in another clinical trial or in period of exclusion from a previous clinical trial

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
parent-proxy QoL chronic cough specific questionnaire (PC-QOL) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France